CLINICAL TRIAL: NCT03212482
Title: Patient-ventilator Asynchrony in Patients With Brain Injury
Status: Completed | Type: Observational
Sponsor: Jian-Xin Zhou (Other)
Responsible Party: Sponsor-Investigator, Jian-Xin Zhou, Doctoral Student Supervisor， chief of the department and Deputy Dean of the hospital, Capital Medical University
Organization: Capital Medical University (Other)
Other Study IDs: KY 2017-028-02
Record Dates: First submitted 2017-07-04; First posted 2017-07-11 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Brain Injuries; Mechanical Ventilation
Keywords: brain-injured patients, patient-ventilator asychrony
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mechanical ventilation is an important support strategy for critically ill patients. It could improve gas exchange, reduce the work of breathing, and improve patient comfort. However, patient-ventilator asynchrony, which defined as a mismatch between the patient and ventilator may obfuscate these goals. Studies have shown that a high incidence of asynchrony (asynchrony index > 10%) is associated with prolonged mechanical ventilation and ICU length of stay and high mortality. So far, there have been only a few studies on the epidemiology of asynchrony in brain-injured patients. Investigators conduct a prospective observational study among brain-injured patients to determine the prevalence, risk factors and outcomes of patient-ventilator asynchrony. Esophageal pressure monitoring, a surrogate for pleural pressure, combined with airway pressure and flow waveforms is used to detect patient-ventilator asynchrony.

ELIGIBILITY:
Inclusion Criteria:

* 1) ]older than 18 years 2) with brain injury in the ICU 3) mechanical ventilated for at least 72 hours

Exclusion Criteria:

* 1) ICU length of stay less than 24 hours 2) enrolled in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with brain injury and receiving MV for at least 72 hours in the intensive care unit, will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
The incidence of patient-ventilator asynchrony in brain-injured patients | Three days
  The incidence of different types of patient-ventilator asynchrony in brain-injured patients.

SECONDARY OUTCOMES:
The risk factors of patient-ventilator asynchrony in brain-injured patients | Three days
  The risk factors of different types of patient-ventilator asynchrony in brain-injured patients

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Study Chair — Acute Brain Injury and Critical Care Research Collaboration, ABC Research Collaboration
Locations (1):
- Jian-Xin Zhou, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Luo XY, He X, Zhou YM, Wang YM, Chen JR, Chen GQ, Li HL, Yang YL, Zhang L, Zhou JX. Patient-ventilator asynchrony in acute brain-injured patients: a prospective observational study. Ann Intensive Care. 2020 Oct 19;10(1):144. doi: 10.1186/s13613-020-00763-8. PMID 33074406